CLINICAL TRIAL: NCT00640835
Title: A Phase 2 Multi-Center Open-label Study to Assess the Safety and Tolerability of a Buprenorphine/Naloxone Film Strip Administered by the Sublingual and Buccal Routes
Brief Title: Safety and Tolerability of Buprenorphine/Naloxone Film Strips
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-07-0001
Record Dates: First submitted 2008-03-14; First posted 2008-03-21 (Estimated); Results first posted 2010-10-26 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2008-10

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual administration (Experimental): Buprenorphine/naloxone film strip administered sublingually
  Interventions: Drug: Buprenorphine/naloxone Film Strip
- Buccal administration (Experimental): Buprenorphine/naloxone film strip administered buccally
  Interventions: Drug: Buprenorphine/naloxone Film Strip

INTERVENTIONS:
Drug: Buprenorphine/naloxone Film Strip — Buprenorphine/naloxone dosed between 4/1 mg to 32/8 mg once a day for 12 weeks by sublingual route
  Arms: Sublingual administration
Drug: Buprenorphine/naloxone Film Strip — Buprenorphine/naloxone dosed between 4/1 mg to 32/8 mg once a day for 12 weeks by buccal route
  Arms: Buccal administration

SUMMARY:
This study will evaluate the safety and tolerability on the oral mucosa of buprenorphine/naloxone film strips administered either sublingually or buccally daily for 12 weeks in opioid dependent individuals who are already on a stable regimen of buprenorphine/naloxone.

DETAILED DESCRIPTION:
Buprenorphine and naloxone soluble film was developed as an alternative dosage form to Suboxone (buprenorphine and naloxone) sublingual tablets and was evaluated for both sublingual and buccal administration. The soluble film dosage is expected to provide the following enhancements and potential advantages over the current Suboxone (buprenorphine and naloxone) product:

* mitigation against unintentional pediatric exposure by providing child-resistant packaging in unit dose format.
* improvement in subject convenience and compliance by ensuring rapid disintegration.
* protection against diversion by providing a dosage form that is very difficult for the subject to remove from the sublingual or buccal mucosa after administration. This provides assurance to the caregiver that the dose has actually been taken appropriately in a supervised setting.
* provision of a unit dose product format for hospital and institutional use.
* decreased product damage during shipping as compared to Suboxone tablets.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Be 18-to-65 years of age, inclusive.
* Have a diagnosis of opioid dependence by medical history according to DSM-IV-TR criteria.
* Be on stable dose of 4 to 32 mg (expressed as the buprenorphine component)daily of Suboxone for at least 30 days.
* If female, have a negative pregnancy test during screening and agree to use an acceptable method of birth control which may include:

Exclusion Criteria:

Subjects must not:

* Have participated in an experimental drug or device study within the last 30 days.
* If female, be breast feeding or lactating.
* Have any medical condition that in the opinion of the physician investigator would preclude the subject from completing the study.
* Have a clinically significant abnormal finding (in the opinion of the Investigator) on oral cavity exam (e.g., active mouth ulcers).
* Have any piercing of the tongue or mouth within 30 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R. Jasinski, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Parkway Medical Center, Birmingham, Alabama
  - Winston Technology Research LLC, Haleyville, Alabama
  - Beeches Family Medicine, Jacksonville Beach, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment commenced 02/28/08 and was completed 04/15/08. All sites were medical clinics.
Pre-assignment Details: Subjects were required to be on a stabilized dose of buprenorphine and naloxone for at least 30 days prior to study drug administration, either during the screening period, or as part of routine medical treatment during the previous 30 days.
Period: Overall Study
Arm/Group | Buprenorphine/Naloxone Film Strip Administered Sublingually | Buprenorphine/Naloxone Film Strip Administered Buccally
Started | 194 | 188
Completed | 118 | 131
Not Completed | 76 | 57
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 12 | 14
Not completed — Physician Decision | 10 | 14
Not completed — Sponsor's Decision | 11 | 7
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 17 | 13
Not completed — Other Reason | 19 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Naloxone Film Strip Administered Sublingually | Buprenorphine/Naloxone Film Strip Administered Buccally | Total
Number analyzed (Participants) | 194 | 188 | 382
Age Continuous [Mean (Standard Deviation); unit: years] | 36.1 (10.19) | 36.7 (10.09) | 36.4 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 142
  Male | 124 | 116 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 194 | 188 | 382
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 192 | 187 | 379
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 194 | 188 | 382
Age Categorical [Number; unit: Participants] — The age categories used for this study were slightly different than the standard values and are reflected as reported in the study.
  Participants
    <21 | 4 | 0 | 4
    21 - 35 | 102 | 99 | 201
    36 - 50 | 71 | 67 | 138
    >50 | 17 | 22 | 39
Severity Grading of Oral Mucosa [Number; unit: Participants] — Safety and tolerability were evaluated at baseline by oral cavity examination. Oral mucosa was graded as follows:
  Grade 0: Normal mucosa Grade 1: Localized mucosal erythema and/or irritation without ulceration Grade 2: Erythema and/or irritation and induration without ulceration Grade 3: Ulceration, with or without any other combination of signs
  Participants
    Grade 0 | 192 | 185 | 377
    Grade 1 | 2 | 1 | 3
    Grade 2 | 0 | 1 | 1
    Grade 3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events Associated With the Oral Cavity.
Description: Safety and tolerability were evaluated during the 12-week Treatment Phase by oral cavity examination and assessment. Oral mucosa was graded as follows:
  Grade 0: Normal mucosa Grade 1: Localized mucosal erythema and/or irritation without ulceration Grade 2: Erythema and/or irritation and induration without ulceration Grade 3: Ulceration, with or without any other combination of signs
Time Frame: 12 weeks
Population: The population was defined as all subjects who received at least a single dose of study drug and was the only population considered in the analysis plan. Missing data values were not imputed.
Measure: Number; unit: Participants
Arm/Group | Buprenorphine/Naloxone Film Strip Administered Sublingually | Buprenorphine/Naloxone Film Strip Administered Buccally
Number analyzed (Participants) | 194 | 188
Participants | 11 | 16

2. Primary Outcome: Number of Subjects With Mild, Moderate or Severe Treatment-emergent Adverse Events Associated With the Oral Cavity
Description: Safety and tolerability were evaluated during the 12-week Treatment Phase by oral cavity examination and assessment.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Buprenorphine/Naloxone Film Strip Administered Sublingually | Buprenorphine/Naloxone Film Strip Administered Buccally
Number analyzed (Participants) | 194 | 188
Participants
  Mild | 9 | 12
  Moderate | 2 | 3
  Severe | 0 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Buprenorphine/Naloxone Film Strip Administered Sublingually | Buprenorphine/Naloxone Film Strip Administered Buccally
Serious Adverse Events (participants affected / at risk) | 4/194 | 2/188
Other Adverse Events (participants affected / at risk) | 11/194 | 16/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone Film Strip Administered Sublingually (N=194) | Buprenorphine/Naloxone Film Strip Administered Buccally (N=188)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine/Naloxone Film Strip Administered Sublingually (N=194) | Buprenorphine/Naloxone Film Strip Administered Buccally (N=188)
Oral mucosal erythema (Gastrointestinal disorders) | 2 | 6
Toothache (Gastrointestinal disorders) | 2 | 4
Sinusitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.